CLINICAL TRIAL: NCT02402036
Title: Regorafenib in Metastatic Colorectal Cancer: An Exploratory Biomarker Study
Brief Title: A Biomarker Study in Patients Getting Regorafenib for Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-0133
Record Dates: First submitted 2015-02-04; First posted 2015-03-30 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2017-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib (Experimental): Regorafenib 120 mg orally daily for 21 days out of a 28 day cycle
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib orally for 21 days every 28 day cycle
  Other Names: Stivarga

SUMMARY:
This is an exploratory biomarker study. Patients with metastatic colorectal cancer will receive regorafenib, which is FDA approved in this setting, on day 1-21 of every consecutive 28 day cycle. Patients will be asked to undergo tumor biopsy at baseline and 2 weeks after starting regorafenib. Peripheral blood samples will be collected at baseline 2 weeks after starting regorafenib, after initiation of cycle 3, and every 4 weeks thereafter.

DETAILED DESCRIPTION:
Tumor tissue collected at baseline and 2 weeks after starting regorafenib will be analyzed for phosphoproteins and RNA. Peripheral blood samples will be collected and banked for protein, miRNA, and mutated DNA analysis.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer suitable for regorafenib treatment
* Life expectancy of at least 12 weeks
* Able to understand and willing to sign written informed consent form
* Adequate bone marrow, liver, and renal function
* Glomerular filtration rate >/= 60 according to the Modified Diet in Renal Disease abbreviated formula
* Women of childbearing potential must have a negative serum pregnancy test
* Subject able to swallow and retain oral medication

Exclusion Criteria:

* Previous assignment to treatment in this study
* Uncontrolled hypertension
* Active or clinically significant cardiac disease
* Evidence or history of Bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding even Grade 3 or higher within 4 weeks prior to start of study medication
* Subjects with thrombotic, embolic, venous or arterial events
* Subjects with any previously untreated or concurrent cancer
* Pheochromocytoma
* Known history of human immunodeficiency virus infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Ongoing infection Grade 2 or higher
* Symptomatic metastatic brain or meningeal tumors
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Renal failure requiring dialysis
* Dehydration Grade 1 or higher
* Seizure disorder requiring medication
* Persistent proteinuria Grade 3 or higher
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise
* History of organ allograft including corneal transplant
* Known or suspected allergy or hypersensitivity to the study drug
* Any malabsorption condition
* Women who are pregnancy or breast-feeding
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Concurrent anticancer therapy
* Concurrent use of another investigational drug or device therapy during or within 4 weeks of trial entry
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
* Therapeutic anticoagulation with Vitamin-K antagonists or with heparins and heparinoids
* Use of any herbal remedy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Weinberg BA, Hartley ML, Salem ME. Precision Medicine in Metastatic Colorectal Cancer: Relevant Carcinogenic Pathways and Targets-PART 2: Approaches Beyond First-Line Therapy, and Novel Biologic Agents Under Investigation. Oncology (Williston Park). 2017 Jul 15;31(7):573-80. PMID 28712102

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regorafenib
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 2
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Serum microRNA Quantification
Description: Serum microRNAs will be quantified using miScript MiRNA PCR arrays
Time Frame: 2 years
Population: Due to issues with recruitment and the principal investigator leaving the institution, no analysis of the collected samples was performed.
Arm/Group | Regorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from the time they signed the informed consent until study completion up to 1 year of treatment and safety follow-up. The period of collection depended on the length of the treatment period.
Arm/Group | Regorafenib
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (N=10)
Abdominal Pain (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hyponatremia (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (N=10)
Abdominal Pain (General disorders) | 5 (7)
Alkaline phosphatase increased (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 3 (5)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Renal and urinary disorders) | 1 (1)
Elevated total bilirrubin (Hepatobiliary disorders) | 2 (3)
High Neutrophils (Immune system disorders) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 4 (7)
Hyponatremia (General disorders) | 2 (3)
PT increased (Blood and lymphatic system disorders) | 1 (1)
WBC increased (Immune system disorders) | 1 (1)
Alanine aminotransferase increased (Hepatobiliary disorders) | 2 (3)
Fatigue (General disorders) | 6 (7)
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 5 (8)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hoarseness (General disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Lymphocyte count decreased (Immune system disorders) | 1 (1)
Nasal bleed (Blood and lymphatic system disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Pain (General disorders) | 3 (6)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth development disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT02402036/Prot_SAP_000.pdf